CLINICAL TRIAL: NCT04004520
Title: Feasibility of Collecting Stress Biomarkers Among Youth Experiencing Homelessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018H0322
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Stress, Physiological
Keywords: stress; cortisol; alpha-amylase; homelessness; biomarkers; virtual reality; meditation
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality with Meditation (Experimental): Participants will receive a virtual reality and audio guided mindfulness meditation program available at (https://guidedmeditationvr.com/)
  Interventions: Behavioral: Virtual Reality with Meditation
- Virtual Reality Control (Other): Participants will receive a virtual reality of historic photographs and written narratives program (https://lookingglassvr.com/)
  Interventions: Behavioral: Virtual reality Control
- Audio Control (Other): Participants will receive an online audio-only guided mindfulness meditation available at (https://www.uclahealth.org/marc/mindful-meditations).
  Interventions: Behavioral: Audio Control

INTERVENTIONS:
Behavioral: Virtual Reality with Meditation — The Guided Meditation Virtual Reality is a mindfulness meditation app provided on a virtual reality platform that includes a 10 minute audio meditation for relaxation along with a 3D visualization of natural settings (e.g. forest, beach, mountain).
  Other Names: Guided Meditation Virtual Reality
  Arms: Virtual Reality with Meditation
Behavioral: Audio Control — The UCLA Mindful App is an audio only mindfulness meditation for relaxation called Breath, Sound, Body Meditation that is 12 minutes in length.
  Other Names: UCLA Mindful App
  Arms: Audio Control
Behavioral: Virtual reality Control — The Looking Glass Virtual Reality is a stereographic 3D photo viewer provided on a virtual reality platform featuring photos from around the world dating back to approximately a century ago that participants will view for 10 minutes.
  Other Names: Looking Glass Virtual Reality
  Arms: Virtual Reality Control

SUMMARY:
The study will examine changes in acute stress (biological and psychological) via salivary cortisol and alpha amylase levels as well as survey measures of self-reported anxiety in response to either (a) a free online guided mindfulness meditation available at (https://www.uclahealth.org/marc/mindful-meditations); (b) a guided mindfulness meditation via virtual reality (https://guidedmeditationvr.com/) or (c) a virtual reality platform of historic photographs and written narratives (https://lookingglassvr.com/). Participants will also complete an interviewer administered survey to measure sociodemographic factors, mental and physical health status, substance use, and medication use and provide a hair sample to measure cortisol.

DETAILED DESCRIPTION:
Homeless youth experience many daily stressors, including hunger, poor sleep, harassment, and violence. Many also have been victims of child abuse and/or neglect, witnessed family and/or community violence, and/or lived in foster care prior to leaving the home setting - exposures labeled as adverse childhood experiences known to increase the risk for poor physical and mental health. Because homeless youth are often disconnected from families, friends and institutions (e.g. health care, schools, jobs), they are at greater risk for "toxic stress" resulting in impaired biological stress responses with high or low levels of the stress hormone, cortisol, and increased inflammation in the cells of the body. High levels of inflammation are associated with sickness behavior syndrome (e.g. fatigue), depression, and suicidal thoughts, which may lead youth to engage in risky behaviors (e.g. substance use, HIV risk behaviors) in an attempt to reduce symptoms. However, few studies have collected biological measures of stress among homeless youth despite prior research linking exposure to violence and trauma to impaired biological stress responses in the general population. Because homeless youth experience a greater number of adverse exposures and with higher levels of severity on a daily basis and across their lifetime than youth in the general population, our lack of understanding of the biological impact that these exposures have on homeless youths' physical and mental health in the short-term as well as across their life span limits understanding of which youth are most vulnerable to poor outcomes. This study's purpose is to test the feasibility of collecting acute and chronic stress response biomarkers in homeless youth for use with future planned research. The study will also assess changes in acute stress (biological and psychological) via salivary cortisol and alpha amylase levels as well as survey measures of self-reported anxiety in response to either (a) a free online guided mindfulness meditation available at (https://www.uclahealth.org/marc/mindful-meditations); (b) a guided mindfulness meditation via virtual reality (https://guidedmeditationvr.com/) or (c) a virtual reality platform of historic photographs and written narratives (https://lookingglassvr.com/). Participants will also complete an interviewer administered survey to measure sociodemographic factors, mental and physical health status, substance use, and medication use and provide a hair sample to measure cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 24 years
* Meets the criteria for homelessness as defined by the federal McKinney-Vento Act as "lacking a fixed, regular, stable, and adequate nighttime residence" and includes "living in a publicly or privately operated shelter designed to provide temporary living accommodations, or a public or private place not designed for, or ordinarily used as, regular sleeping accommodations for human beings"
* speaks and understands the English language

Exclusion Criteria:

* 17 years and younger
* 25 years and older
* non-English speakers

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Change in Stress Reactivity | Baseline, 5 minutes, 20 minutes, 35 minutes
  Participant gives the first saliva sample at arrival, then the second saliva sample 5 minutes after arrival prior to the intervention. The intervention is administered (approximately 10-15 minutes in length). The participant will give the third saliva sample immediately after the intervention and then a fourth saliva sample 15 minutes after the intervention.

SECONDARY OUTCOMES:
Change in Self-reported Anxiety as measured by the Spielberger State-Trait Anxiety Inventory | 5 minutes, 35 minutes
  The Spielberger State-Trait Anxiety Inventory survey which has six-item short-form of the state(STAI: Y-6 score.
  To calculate the total STAI score (range 20 - 80):
  * reverse scoring of the positive items (calm, relaxed, content) so 1=4, 2=3, 3=2 and 4=1;
  * sum all six scores;
  * multiply total score by 20/6;
  * refer to Spielberger's manuals to interpret scores (a 'normal' score is approx. 34 - 36)
  Participant will complete the survey 5 minutes prior to the intervention and then 15 minutes after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi L Ford, PhD, Study Chair — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chavez LJ, Kelleher K, Slesnick N, Holowacz E, Luthy E, Moore L, Ford J. Virtual Reality Meditation Among Youth Experiencing Homelessness: Pilot Randomized Controlled Trial of Feasibility. JMIR Ment Health. 2020 Sep 24;7(9):e18244. doi: 10.2196/18244. PMID 32969834
- See also: Guided Meditation VR — https://guidedmeditationvr.com
- See also: Looking Glass VR — https://lookingglassvr.com/
- See also: UCLA Mindful Meditation — https://www.uclahealth.org/marc/mindful-meditations